CLINICAL TRIAL: NCT00868647
Title: Radiofrequency Ablation (RFA) Of Tumors Acquired In Childhood: A Phase II Study
Brief Title: Radiofrequency Ablation (RFA) Of Tumors Acquired In Childhood
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Fredric A. Hoffer MD FAAP, FSIR, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RFAII
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Last update posted 2009-09-01 (Estimated); Status verified 2009-08

CONDITIONS: Neoplasms, Benign; Neoplasms, Malignant
MeSH Terms: conditions — Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiofrequency Ablation (Other)
  Interventions: Procedure: Radiofrequency ablation (RFA)

INTERVENTIONS:
Procedure: Radiofrequency ablation (RFA) — Radiofrequency tumor ablation (RFA) is an imaging guided percutaneous or intra-operative procedure that uses a probe on the end of a sharp needle that is inserted directly into the tumor. The tumor is ablated by heating the probe (using electrical current alternating at radio frequency) which raises the temperature of the tumor potentially causing irreversible cell death.

SUMMARY:
This is a single-center, Phase II study including only patients on whom a decision to conduct radiofrequency ablation (RFA) has already been made. The primary objective of this study assess if quality of life was improved by RFA as assessed at baseline, 3 and potentially 6 and 12 months following RFA for the benign lesions.

RFA is an imaging guided percutaneous or intra-operative procedure that uses a probe on the end of a sharp needle that is inserted directly into the tumor. The tumor is ablated by heating the probe (using an electrical current alternating at radio frequency) which raises the temperature of the tumor potentially causing irreversible cell death.

RF ablation is an alternative for local tumor control when other treatments (surgery, radiotherapy or chemotherapy) are not feasible (less effective or at higher risk). Thermal ablation at times is the only remaining alternative for patient cure, prolonged survival or palliation. Cryotherapy, and microwave, laser and focused ultrasound are alternative thermal ablation techniques used in adults but there has been no experience in children with these alternative methods.

To be eligible for this study, patients must have acquired lesions at < 21 years of age (central nervous system lesions are excluded from this study). Study participants will have the RFA procedure performed at Seattle Children's and will have follow-up evaluations at various time points post-RFA.

ELIGIBILITY:
Inclusion Criteria:

* Lesion acquired in childhood (at <21 years of age)
* Any lesion location except CNS
* Any malignant tumor or metastasis
* Any benign lesion (e.g. desmoids, venous or lymphatic vascular anomalies, aneurysmal bone cysts, osteoid osteoma, tongue hypertrophy, or painful neuropathy)
* Patients with malignant disease have had histologic confirmation of disease at initial diagnosis.
* ≥ 90 day life expectancy
* Potential benefit of RFA outweighs risk as determined by PI
* Other local tumor control measures are not recommended for malignant lesion based on review in multidisciplinary team conference or the patient refuses recommended local tumor control measures
* The patient is not expected to become short of breath at rest after RFA (forced vital capacity ≥33% of normal by pulmonary function tests) if pulmonary RFA is considered

Exclusion Criteria:

* Patients with uncontrolled infection.
* Patients with co-morbidities affecting inclusion criteria above.
* Patients who are pregnant and/or breastfeeding.
* Patients who had a change in chemotherapy within one month before RFA
* Patients who have planned change in chemotherapy and/or radiation therapy (to same site as RFA) interventions within the first three months following RFA.
* Patients should not be considered for pulmonary RFA if they have poorly compliant lungs (recently required mechanical ventilation) or require supplemental oxygen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-06; Primary Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Assess if quality of life was improved by RFA for the benign lesions | baseline, 3 months and potentially 6 and 12 months following RFA

SECONDARY OUTCOMES:
Assess the response to RF ablative therapy by pain relief from painful benign or malignant lesions. | baseline, 3 months and potentially 6 and 12 months following RFA
Evaluate the rate of short-term ablation of benign lesions produced by RFA | baseline, 3 months and potentially 6 and 12 months following RFA
Assess toxicity related to all RFA procedures using the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | within 3 months (potentially 6-12 months) following RFA
Assess the response to RFA by malignant tumor markers (e.g. AFP) | 1, 3, 6, and 12 months following RFA
Assess if quality of life was improved by RFA for patients with malignant lesions | baseline, 3, 6 and 12 months
Evaluate the proportion of malignant lesions that show short-term ablation produced by RFA. | 3 months post Radiofrequency Ablation (RFA), as compared to 1 month post RFA imaging
Determine the rate of durable ablation in malignant lesions that achieve short-term ablation by RFA | 12 months post RFA
Assess the time to malignant tumor progression (as defined by RECIST) of lesions treated with RFA | 1, 3, 6, and 12 months post RFA

CONTACTS AND LOCATIONS:
Overall Officials: Fredric A Hoffer, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States